CLINICAL TRIAL: NCT06016842
Title: A Phase III Randomised, Parallel-Group, Double-Blind, Placebo-Controlled, Two-Arm Study to Evaluate the Efficacy and Safety of Elafibranor 80 mg on Long-Term Clinical Outcomes in Adult Participants With Primary Biliary Cholangitis (PBC)
Brief Title: A Long-Term Study of Elafibranor in Adult Participants With Primary Biliary Cholangitis
Acronym: ELFIDENCE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIN-60190-454; 2023-505251-43-00 (EU CTIS Number)
Record Dates: First submitted 2023-08-22; First posted 2023-08-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Primary Biliary Cholangitis (PBC)
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elafibranor 80 mg (Experimental): Participants will take 1 tablet of elafibranor 80 mg per day orally before breakfast with a glass of water at approximately the same time each morning.
  Interventions: Drug: Elafibranor
- Placebo (Placebo Comparator): Participants will take 1 placebo tablet per day orally (matching the 80 mg elafibranor sized tablet) before breakfast with a glass of water at approximately the same time each morning.
  Interventions: Other: Matched 80 mg placebo

INTERVENTIONS:
Drug: Elafibranor — Duration: up to an estimated 42-month (3.5-year) double-blind treatment period during which elafibranor 80 mg tablet will be administered once daily
  Arms: Elafibranor 80 mg
Other: Matched 80 mg placebo — Duration: up to an estimated 42-month (3.5-year) double-blind treatment period during which matching placebo tablet will be administered once daily
  Arms: Placebo

SUMMARY:
The participants of this study will have confirmed Primary Biliary Cholangitis (PBC) and cirrhosis (scarring of the liver).

PBC is a slowly progressive disease, characterised by damage to the bile ducts in the liver, leading to a build-up of bile acids which causes further damage.

The liver damage in PBC may lead to cirrhosis. PBC may also be associated with multiple symptoms. Many patients with PBC may require liver transplant or may die if the disease progresses and a liver transplant is not done.

This study will compare a daily dose of elafibranor (the study drug) to a daily dose of placebo (a dummy treatment) and will last up to 3.5 years for each participant.

The main aim of this study is to determine if elafibranor is better than placebo in preventing clinical outcome events showing disease worsening (including progression of disease leading to liver transplant or death).

This study will also study the safety of long-term treatment with elafibranor, as well as the impact on symptoms such as itching and tiredness.

ELIGIBILITY:
Inclusion Criteria :

* Male or female participants must be ≥18 years of age at the time of signing the informed consent.
* Participants with a definite or probable diagnosis of primary biliary cholangitis (PBC)
* Participants with cirrhosis at SV1. • Participants must be Child Pugh A or Child Pugh B.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria :

* History or presence of other concomitant liver disease including but not limited to:

  * i) Primary sclerosing cholangitis (PSC).
  * ii) Autoimmune hepatitis (AIH) by simplified Diagnostic Criteria of the International Autoimmune Hepatitis Group (IAIHG) ≥6, or if treated for an overlap of PBC with AIH, or if there is clinical suspicion and evidence of overlap AIH features, that cannot be explained alone by insufficient response to UDCA.
  * iii) Positive hepatitis B surface antigen (HBsAg). Participants with negative HBsAg and positive hepatitis B core antibody (HBcAb) may be eligible if hepatitis B virus deoxyribonucleic acid (HBV DNA) is negative.
  * iv) Hepatitis C virus (HCV) infection defined by positive anti-HCV antibody and positive HCV ribonucleic acid (RNA) (Note: Participants with positive anti-HCV antibody due to previously treated HCV infection, may be enrolled if a confirmatory HCV RNA is undetectable and sustained viral response has been documented).
  * v) Alcohol-associated liver disease (ALD).
  * vi) Nonalcoholic steatohepatitis (NASH).
  * vii) Other chronic liver diseases, such as alpha-1 antitrypsin deficiency.
* History or presence of clinically significant hepatic decompensation, including:

  * i) History of liver transplantation, current placement on a liver transplant list, current model for end-stage liver disease including (MELD) 3.0 score >12 due to hepatic impairment.
  * ii) Evidence of complications of cirrhosis, including hepatic decompensation or evidence of significant portal hypertension complications including presence of uncontrolled ascites; history of variceal bleeding or related interventions (e.g. variceal banding, or transjugular intrahepatic portosystemic shunt placement); presence of hepatic encephalopathy Grade 2 or higher per West-Haven criteria; history or presence of spontaneous bacterial peritonitis. Note: participants with low-risk varices (Grade I) without history of bleeding or other treatment may be eligible to enrol.
  * iii) Hepatorenal syndrome (HRS) (type I or II ). • vi) Hospitalisation for liver-related complication within 12 weeks prior to SV1.
* Known history of human immunodeficiency virus (HIV) infection or having a positive confirmatory test for HIV type 1 or 2.
* Medical conditions that may cause non-hepatic increases in ALP (e.g. Paget's disease).
* Evidence of any other unstable or untreated clinically significant immunological, endocrine, hematologic, gastrointestinal, neurological, or psychiatric disease as evaluated by the investigator; other clinically significant conditions that are not well controlled.
* Non-hepatic medical conditions that may diminish life expectancy to <2 years, including known cancers.
* History of hepatocellular carcinoma.
* Alpha-fetoprotein (AFP) >20 ng/mL with 4-phase liver computerised tomography (CT) or magnetic resonance imaging (MRI) imaging suggesting presence of hepatocellular carcinoma.
* Known malignancy or history of malignancy within the last 5 years, with the exception of local, successfully treated basal cell carcinoma or in-situ carcinoma of the uterine cervix.
* Administration of the following medications is prohibited during the study, and prior to the study as per the timelines specified below: • i) 3 months prior to screening period: fibrates, seladelpar, glitazones, obeticholic acid, azathioprine, cyclosporine, methotrexate, mycophenolate, pentoxifylline, budesonide and other systemic corticosteroids (parenteral and oral chronic administration only); potentially hepatotoxic drugs (including α-methyl-dopa, sodium valproic acid, isoniazid or nitrofurantoin).
* Participants who are currently participating in, plan to participate in, or have participated in an investigational drug study or medical device study containing active substance within 30 days or 5 half-lives, whichever is longer, prior to the screening period.

  i) If the previous study was for an experimental therapy being studied for potential benefit in PBC, and the potential therapeutic agent was proven to have no beneficial effect in PBC and there are no safety concerns, the participant may enrol after 30 days or 5 half-lives from the last dose of the therapeutic agent, whichever is longer.ii) For therapeutic agents being studied for potential benefit in PBC for which it is still unclear if there may be a potential benefit, participants may enrol after 6 months from the last dose of the therapeutic agent.
* Electrocardiogram (ECG) with QT interval corrected by Fridericia's formula (QTcF) >450 msec in males or QTcF >470 msec in females for participants without bundle branch block. For participants with bundle branch block or other intraventricular conduction delay, a longer QTcF >480 msec would be exclusionary.
* Total bilirubin (TB) >5x ULN
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >5x ULN at SV1
* Creatinine phosphokinase (CPK) >2x ULN.
* Platelet count <50,000/μL
* International normalised ratio (INR) >1.8 in the absence of anticoagulant therapy.
* Estimated glomerular filtration rate (eGFR) <45 mL/min/1.73m2 per the Modification of Diet in Renal Disease (MDRD)-6 Study formula at SV1.
* Significant renal disease, including nephritic syndrome, chronic kidney disease (CKD) (defined as participants with evidence of significantly impaired kidney function or underlying kidney injury).
* For female participants: known current pregnancy, or has a positive serum pregnancy test, or is breastfeeding.
* Participants unwilling or unable to be abstinent from alcohol during the study.
* History of alcohol abuse, or other substance abuse within 1 year prior to SV1.
* Known hypersensitivity to elafibranor or to any of the excipients of the investigational product(s).
* Mental instability or incompetence, such that the validity of informed consent or ability to be compliant with the study is uncertain.
* Any other condition that, in the opinion of the investigator, would interfere with study participation or completion, or would put the participant at risk, including a potential participant assessed as being at high risk of noncompliance with the study.
* Alkaline phosphatase (ALP) ≥10x ULN.
* Albumin <2.8 g/dL due to impaired hepatic function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | From baseline until 4 weeks after the end of treatment (maximum duration of 3.5 years)
  Event-free survival is defined as the time from randomisation to either adjudicated disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Percentage of participants experiencing Treatment Emergent Adverse Events (TEAEs), treatment-related TEAEs, Serious Adverse Events (SAEs), and Adverse Events of Special Interests (AESIs) | From baseline until 4 weeks after the end of treatment (maximum duration of 3.5 years)
  An Adverse event (AE) is any untoward medical occurrence, temporally associated with the use of study intervention, whether or not related to the study intervention. AESIs are AEs that may not be serious but are of special importance to a particular drug or class of drugs.
Percentage of participants developing clinically significant changes in physical examination findings | From baseline until 4 weeks after the end of treatment (maximum duration of 3.5 years)
  Complete physical examination at screening and targeted examination at all other clinical visit timepoints.
Percentage of participants developing clinically significant changes in vital signs | From baseline until 4 weeks after the end of treatment (maximum duration of 3.5 years)
  Percentage of participants with clinically significant changes in Vital Signs will be reported. The clinical significance will be graded by the investigator.
Percentage of participants developing clinically significant changes in Electrocardiogram (ECG) readings. | From baseline until 4 weeks after the end of treatment (maximum duration of 3.5 years)
  Percentage of participants with clinically significant changes in ECG readings will be reported. The clinical significance will be graded by the investigator.
Percentage of participants with clinically significant changes in laboratory parameters (blood chemistry, hematology, coagulation and urinalysis) | From baseline until 4 weeks after the end of treatment (maximum duration of 3.5 years)
  Percentage of participants with clinically significant change in laboratory parameters (blood chemistry, hematology and coagulation) will be reported. The clinical significance will be graded by the investigator.
Change from baseline in Alkaline phosphatase (ALP) | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Change from baseline in Total Bilirubin (TB) | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Percentage of participants with ALP≤ 1.67x ULN and TB≤ ULN | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Percentage of participants with complete biochemical response | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
  Defined as normal levels of TB, ALP, transaminases, albumin, and International normalised ratio (INR)
Percentage of participants with normalisation of TB and ALP | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
  Defined as TB< Upper Limit Normal (ULN) and ALP< ULN
Percentage of participants with stabilisation in TB (i.e. no increase) | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
  Defined as TB< 1x ULN or increase from baseline <0.1x ULN
Percentage of participants with a response based on albumin normalisation | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Change from baseline in liver stiffness measurement (LSM) | At Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
  Assessed by vibration-controlled transient elastography (VCTE) using Fibroscan® on the day of the visit.
Change from baseline in PBC risk scores based in Global PBC Study Group (GLOBE) score | At Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
  The GLOBE score is a validated risk assessment tool providing an estimate of transplant-free survival for patients with PBC. It was developed by the Global PBC Study Group using Cox regression model on over 4,000 patients with PBC. Lower GLOBE score predicts lower risk. It is calculated from the following equation:
  GLOBE score = (0.044378 * age + 0.93982 * LN(total bilirubin/ULN) +(0.335648 * LN(alkaline phosphatase/ULN)) - 2.266708 * albumin /LLN -0.002581 * platelet count per 109/L) + 1.216865
  GLOBE scoring system, which calculation is based on serum values of bilirubin, ALP, albumin and platelet count after 1 year of treatment and age at baseline. A high number is indicative of a worse score.
Change from baseline in PBC risk scores based on United Kingdom (UK)-PBC score. | At Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
  PBC risk score developed by United Kingdom (UK)-PBC Consortium is a scoring system and the calculation is based on laboratory test measurements and upper limits of normal (ULN) for the total bilirubin (BIL12); alanine transaminase or aspartate transaminase (TA12), and alkaline phosphatase (ALP12) after at least 12 months of UDCA, and the laboratory test measurements and lower limits of normal (LLN) for the serum albumin and platelet count in the same timeframe. A high number is indicative of a worse score.
Percentage of participants with LSM ≥15 kPa | At Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
  Assessed by VCTE using Fibroscan®
Change in serum levels of Aspartate aminotransferase (AST) compared to the baseline | At Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Change in serum levels of ALT compared to the baseline | At Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Change in serum levels of Gamma-glutamyl transferase (GGT) compared to the baseline | At Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Change from baseline in hepatic function: Conjugated bilirubin | At Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Change in serum levels of Albumin compared to the baseline | At Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Change from baseline in hepatic function: international normalised ratio (INR) | At Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Change from baseline in hepatic function: fractionated ALP | At Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Percentage of participants with no worsening of LSM | At Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
  Assessed by VCTE using Fibroscan® defined as no increase >2kPa from baseline
Percentage of participants with ALP reduction of 40% | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Percentage of participants with ALP <1.5x ULN, ALP decrease ≥15% and TB ≤ULN | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Percentage of participants with ALP <1.5x ULN, ALP decrease ≥40% and TB ≤ULN | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Percentage of participants with ALP <1.67x ULN, ALP decrease ≥15% and TB ≤ULN | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Percentage of participants with ALP <3x ULN, AST <2x ULN and TB ≤1 mg/dL (Paris I) | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Percentage of participants with ALP ≤1.5x ULN, AST ≤1.5x ULN and TB ≤1 mg/dL (Paris II criteria) | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Percentage of participants with normalisation of abnormal TB | Assessed at Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Percentage of participants with normalisation of abnormal TB and albumin (Rotterdam criteria) | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Percentage of participants with reduction in TB to ≤0.6x ULN in participants with TB >0.6x ULN at baseline | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Change from baseline in lipid parameters: total cholesterol (TC) | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Change from baseline in lipid parameters: high density lipoprotein cholesterol (HDL-C) | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Change from baseline in lipid parameters: calculated very low density lipoprotein cholesterol (VLDL-C) | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Change from baseline in lipid parameters: low density lipoprotein cholesterol (LDL-C) | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Change from baseline in lipid parameters: triglycerides (TG) | At Month 6, Month 12, and every 12 months up to end of treatment (maximum duration of 3.5 years)
Percentage of participants with a response in PBC Worst Itch NRS score | Through 6 months up to end of treatment (maximum duration of 3.5 years)
  Defined as ≥2-point reduction from baseline NRS in participants with a baseline NRS ≥4
Percentage of participants with a response in PBC Worst Itch NRS | Assessed through 6 months up to end of treatment (maximum duration of 3.5 years)
  Defined as ≥3-point reduction from baseline NRS in participants with a baseline NRS ≥4
Change from baseline in 5D-Itch scale | Assessed at every 6 months up to end of treatment (maximum duration of 3.5 years)
  Questionnaire that assesses symptoms in terms of 5 domains: degree, duration, direction, disability and distribution. Participants rate their symptoms over the preceding 2-week period on a 1 to 5 scale, with 5 being the most affected.
Change from baseline in Patient Global Impression of Severity (PGI-S) | Assessed at every 6 months up to end of treatment (maximum duration of 3.5 years)
  A 1-item, 5-point scale designed to assess the participant's impression of disease severity
Patient Global Impression of Change (PGI-C) | Assessed at every 6 months up to end of treatment (maximum duration of 3.5 years)
  A 1-item, 5-point scale designed to assess the participant's impression of change in disease severity since the baseline visit
Change from baseline in Patient Reported Outcome Measurement Information System (PROMIS) Fatigue Short Form 7a | Assessed at every 6 months up to end of treatment (maximum duration of 3.5 years)
  Consists of 7 items that measure both the experience of fatigue and the interference of fatigue on daily activities over the past week. Response options are on a 5-point Likert scale, ranging from 1 to 5. Scores can range from 7 to 35, with higher scores indicating greater fatigue.
Change from baseline in the Epworth Sleepiness Scale (ESS) | Assessed at every 6 months up to end of treatment (maximum duration of 3.5 years)
  Self-administered questionnaire that consists of 8 questions asking to rate how likely it is to fall asleep in different situations commonly encountered in daily life (each question can be scored from 0 to 3 points; '0' indicates no sleepiness, '3' indicates significant sleepiness). It provides a total score which has been shown to relate to the participant's level of daytime sleepiness (total score range 0-24 points).
Change from baseline in PBC-40 score | Assessed at every 6 months up to end of treatment (maximum duration of 3.5 years)
  40-item questionnaire that assesses symptoms across 6 domains: fatigue, emotional and social, cognitive function, general symptoms and itch. Participants respond on a verbal response scale, depending on the section options range from 'never' / 'not at all' / 'strongly disagree' to 'always' / 'very much' / 'strongly agree'. Six items (3/3 in the itch domain, 2/10 in the social domain, and 1/7 in the general symptoms domain) also include a 'does not apply' option. A score for each domain is provided (but a total score is not calculated), with each verbal response scale correlating to a score of 1 to 5 per item (0 to 5 on items with a 'does not apply' option) with 5 being the most affected (greatest burden). The PBC-40 has a 4-week recall period.
Change from baseline in PBC Worst Itch Numeric Rating Scale (NRS) score | Assessed through 6 months up to end of treatment (maximum duration of 3.5 years)
  Self-administered patient-reported outcome questionnaire that measures itch intensity. It asks participants to rate the intensity of their Worst Itch on an 11-point scale ranging from 0 (no itch) to 10 (Worst Itch imaginable): - once daily (24-hour recall period) using the eDiary during the screening and initial 2 years of the study, - at the clinic visits (7-day recall period), from Year 3 onwards
Change from baseline in EuroQol 5-dimensional 5-level questionnaire (EQ-5D-5L) | Assessed at every 6 months up to end of treatment (maximum duration of 3.5 years)
  Self-administered standardised questionnaire that assesses the 5-dimensions of mobility, self-care, usual activities, pain/discomfort, anxiety/depression descriptively (each dimension has 5 levels) and the overall health state via an EQ Visual Analogue Scale (VAS).
Change from baseline in Work Productivity and Activity Impairment General Health (WPAI-GH) | Assessed at every 6 months up to end of treatment (maximum duration of 3.5 years)
  Questionnaire that measures absenteeism, presenteeism as well as the impairments in unpaid activity because of health problem during the past seven days. It consists of 6 questions: 1=currently employed; 2=hours missed because of health problems; 3=hours missed because of other reasons; 4=hours actually worked; 5=degree health affected productivity while working (using a 0 to 10 Visual Analogue Scale (VAS)); 6=degree health affected productivity in regular unpaid activities (VAS).
Time to the first occurrence of each of individual adjudicated clinical outcome events | From baseline until 4 weeks after the end of treatment
  Among: • All-cause mortality • Liver-related mortality • Liver transplant • MELD-3.0 score ≥15 in participants with baseline MELD score ≤12 • Liver decompensation
Area under the plasma concentration-time curve from time 0 to 24 hours: AUC0-24 | At Day 1/Baseline, Month 6 and Month 12 (during a dosing period of 24 hours)
Maximum (peak) plasma drug concentration: Cmax | At Day 1/Baseline, Month 6 and Month 12 (during a dosing period of 24 hours)
Time to reach maximum (peak) plasma concentration following drug administration): Tmax | At Day 1/Baseline, Month 6 and Month 12 (during a dosing period of 24 hours)
Apparent clearance of drug from plasma (CL) | At Day 1/Baseline, Month 6 and Month 12 (during a dosing period of 24 hours)
Apparent volume of distribution (VZ) | At Day 1/Baseline, Month 6 and Month 12 (during a dosing period of 24 hours)
Change from baseline in model for end-stage liver disease (MELD) 3.0 score | From screening until end of treatment (maximum duration of 3.5 years)
  The MELD 3.0 score is calculated from parameters (sex, creatinine, bilirubin, INR, sodium and albumin) where a high score indicates a greater risk of needing a liver transplant.
Change from baseline in Child Pugh grade | From screening until end of treatment (maximum duration of 3.5 years)
  Child Pugh grade is calculated using bilirubin, albumin, INR, ascites and encephalopathy.
  A high grade is indicative of worse liver disease.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (171):
- United States (40):
  - Arizona Liver Health, Tucson, Arizona
  - Arkansas Diagnostic Center, PA, Little Rock, Arkansas
  - Southern California Research Center, Coronado, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - GastroIntestinal BioSciences, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - South Denver Gastroenterology, P.C., Englewood, Colorado
  - Rocky Mountain Gastroenterology, Littleton, Colorado
  - University Of Miami School Of Medicine, Center For Liver Diseases, Miami, Florida
  - Bolanos Clinical Research, Pembroke Pines, Florida
  - International Center for Research, Tampa, Florida
  - University of Kansas Medical Center (KUMC) - University of Kansas Liver Center - Hepatology Clinic, Kansas City, Kansas
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - Huron Gastroenterology Associates - Center for Digestive Care, Ypsilanti, Michigan
  - Southwest Gastroenterology Associates, PC (SWGA), Albuquerque, New Mexico
  - NYU Langone Gastroenterology and Hepatology Associates, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Gastroenterology Center of the Midsouth, Cordova, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - American Research Corporation, Austin, Texas
  - Rush University Medical Center - University Cardiovascular Surgeons, Dallas, Texas
  - Liver Center of Texas, Dallas, Texas
  - Methodist Transplant Physicians, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor Scott & White All Saints Medical Center - Forth Worth, Fort Worth, Texas
  - Liver Associates of Texas, Houston, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - Gastro health & Nutrition, Katy, Texas
  - American Research Corporation at The Texas Liver Institute, San Antonio, Texas
  - Impact Research Tx, Waco, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Inc, Richmond, Virginia
  - Virginia Commonwealth University Medical Center - West Hospital, Richmond, Virginia
  - Medstar Georgetown Transplant Institute University Hospital (MGUH), Columbia, Washington
  - Velocity Clinical Research at Liver Institute Northwest, Seattle, Washington
- Argentina (8):
  - DIM Centro Medico, Buenos Aires
  - Fundacion Respirar (Centro Medico Dra. De Salvo) - Instituto Argentino de Investigaciones Clinicas (IAIC) S.R.L, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Centro Medico Colon, Córdoba
  - Hospital Espanol de Mendoza, Mendoza
  - Hospital Universitario Austral, Pilar
  - Hospital El Cruce, San Juan Bautista
- Australia (6):
  - Sunshine Coast University Hospital, Birtinya
  - Footscray Hospital, Western Health, Footscray
  - Nepean Clinical School, Kingswood
  - Monash University - Monash Health -Monash Medical Centre, Melbourne
  - St George Hospital, Sydney
  - Westmead Hospital, Westmead
- Belgium (4):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Ziekenhuis Oost-Limburg, Genk
  - Gent University Hospital, Ghent
  - Algemeen Ziekenhuis Delta, Roeselare
- Brazil (7):
  - NUPEC Cardio, Belo Horizonte
  - Universidade Federal de Goias, Goiânia
  - Hospital de Clinicas de Porto Alegre (HCPA), Porto Alegre
  - Instituto D'Or de Pesquisa e Ensino - Hospital Aliança, Salvador
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
  - Hospital de Base - Centro Integrado de Pesquisa ( CIP ), São Paulo
  - Universidade Estadual Paulista Julio De Mesquita Filho (UNESP) Hospital das Clinicas Faculdade de Medicina de Botucatu (HCFMB), São Paulo
- Bulgaria (3):
  - Diagnostic-Consultative Center Aleksandrovska EOOD, Sofia
  - Tokuda Hospital, Dept. of Internal Medicine, Sofia
  - University Hospital City Clinic Cancer Center, Sofia
- Canada (2):
  - University of Alberta - Faculty of Medicine & Dentistry - The Centre of Excellence for Gastrointestinal Inflammation and Immunity Research (CEGIIR), Edmonton
  - University Health Network (UHN) - Toronto General Hospital (TGH) - Toronto General Research Institute (TGRI), Toronto
- Chile (6):
  - Universidad De Los Andes, Las Condes
  - Centro de Estudios Clinicos e Investigaciones Medicas (CECIM), Santiago
  - Enroll SpA, Santiago
  - Hospital Clinico de la Pontificia Universidad Catolica de Chile, Santiago
  - University of Chile Clinical Hospital (Hospital Clinico de la Universidad de Chile), Santiago
  - Centro Medico Cedid - Centro de Diagnostico Digestivo, Viña del Mar
- Czechia (5):
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Krajska Nemocnice Liberec, Liberec
  - Artroscan, Ostrava
  - Research Site s.r.o., Pilsen
  - Institute for Clinical and Experimental Medicine - IKEM, Prague
- Bispebjerg Hospital, Copenhagen, Denmark
- France (8):
  - Centre Hospitalier Regional Universitaire de Lille - Hopital Claude Huriez, Lille
  - Hospices Civils de Lyon (HCL) - Hopital de la Croix-Rousse, Lyon
  - Hopital Saint Joseph - Marseille, Marseille
  - CHU de Nice, Hopital de l'Archet, Nice
  - Assistance Publique - Hopitaux de Paris (AP-HP) - Hopital Universitaire Pitie Salpetriere (Hopital Pitie-Salpetriere), Paris
  - CHU Poitiers, Poitiers
  - Clinique Pasteur, Toulouse
  - Hopital Paul-Brousse - APHP, Villejuif
- Greece (4):
  - Agios Savvas Regional Cancer Hospital, Athens
  - General Hospital of Athens Laiko, Athens
  - General Oncological Hospital of Kifisia Oi Agioi Anargyroi, Athens
  - GeneIppokratio General Hospital of Thessaloniki, Thessaloniki
- Hungary (3):
  - Central Hospital of Northern Pest - Military Hospital, Budapest
  - Kenezy County Hospital, Debrecen
  - Szegedi Tudomanyegyetem AOK, I. sz Belgyogyaszati Klinika, Szeged
- Israel (7):
  - Institute of Gastroenterology and Liver Diseases - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus (RHCC), Haifa
  - Hadassah University Hospital (HUH) - Ein-Kerem, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Galilee Medical Center, ZIV Medical Center, Nahariya
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center - Beilinson Hospital - Liver Institute, Petah Tikva
- Italy (8):
  - Azienda Ospedaliero Universitaria Modena, Modena
  - Ospedale San Gerardo, Monza
  - Azienda Ospedaliero Universitaria Federico II di Napoli, Naples
  - Azienda Ospedaliera di Padova - U.O.C. di Gastroenterologia, Padua
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas, Kaunas
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Mexico (3):
  - Centro de Investigacion Medico Biologica y Terapia Avanzada, Jalisco
  - Centro de Investigacion y Gastroenterologia SC, Mexico City
  - Medical Care & Research, Yucatán
- New Zealand (2):
  - Canterbury District Health Board, Christchurch
  - Waikato Hospital, Hamilton
- Poland (12):
  - NZOZ Twoje Zdrowie EL Sp. z o.o., Elblag
  - Uniwersyteckie Centrum Kliniczne im. Prof. K. Gibinskiego Slaskiego Uniwersytetu Medycznego, Katowice
  - Krakowskie Centrum Medyczne Sp.z.o.o - FutureMeds, Krakow
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Medrise Sp. z o.o., Lublin
  - Krakowskie Centrum Medyczne Sp.z.o.o. - FutureMeds, Małogoskie
  - Centrum Medyczne Medyk Sp. z o.o. Sp. K., Rzeszów
  - Niepubliczny Zaklad Opieki Zdrowotnej (NZOZ) - Poliklinika Doktora Bessera, Sosnowiec
  - FutureMeds Warszawa Centrum, Warsaw
  - FutureMeds sp. z o. o, Wroclaw
  - Nzoz Centrum BadanKlinicznych, Wroclaw
  - PlanetMed Sp. z o.o., Wroclaw
- Romania (5):
  - Centrul Pentru Studiul Metabolismului, Bucharest
  - Sana S.R.L, Bucharest
  - Spital Clinic Dr I Cantacuzino, Bucharest
  - Cluj County Clinical Emergency Hospital, Cluj-Napoca
  - Gastromedica Srl, Iași
- Slovakia (3):
  - Gastroenterological Centre Thalion, Bratislava
  - Univerzitna nemocnica L. Pasteura Kosice, Košice
  - Fakultna nemocnica Nitra, Nitra
- South Korea (19):
  - Pusan National University Hospital (PNUH), Busan
  - Keimyung University Dongsan Hospital, Daegu
  - The Catholic University of Korea Daejeon St.Mary's Hospital, Daejeon
  - Inje University Ilsan Paik Hospital, Goyang-si
  - Korea University Ansan Hospital, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Kyungpook National University Hospital (KNUH), Junggu
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Chung-Ang University Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Bundang Hospital (SNUBH), Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Uijeongbu St. Mary's Hospital, Uijeongbu-si
- Spain (13):
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Clinica Universidad Navarra-Sede Madrid, Madrid
  - Hospital General Universitario Gregorio Maranon (HGUGM), Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital De Montecelo, Pontevedra
  - Institut d Investigacio i Innovacio Parc Tauli, Hospital Universitari Parc Tauli, Sabadell
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/